CLINICAL TRIAL: NCT06033534
Title: Safety and Efficacy Evaluation of the STIMULAN Device for the Slow Release of Antibiotics in Exposed Fractures in the Prevention of Infections, and Creation of an AI Predictive Model for the Risk of Infections: a Prospective, Monocentric, Randomized, Blind Study
Brief Title: Evaluation of STIMULAN Device and AI Model in Preventing Fracture Infections
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Università Vita-Salute San Raffaele (Other)
Responsible Party: Principal Investigator, Professor Giacomo Placella, Associate Professor, Università Vita-Salute San Raffaele
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ATinFE
Record Dates: First submitted 2023-09-04; First posted 2023-09-13 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Open Fracture
MeSH Terms: conditions — Fractures, Open

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STIMULAN DEVICE USED (Experimental): Patients allocated to this arm will receive an extended-release antibiotic device, STIMULAN, as a prophylactic measure against bacterial infection post-fracture repair surgery. The device is designed to release antibiotics in a controlled manner over a specified period of time.
  Interventions: Device: STIMULAN
- STIMULAN DEVICE NOT USED (No Intervention): Patients in this arm will undergo the surgical repair of their open fracture but will not receive any antibiotic device for prophylaxis against bacterial infections.

INTERVENTIONS:
Device: STIMULAN — Procedures:
  Surgical repair of the open fracture, as per standard-of-care guidelines. Insertion of the STIMULAN device at the site of the fracture. Standard post-operative care, including monitoring of inflammatory markers and clinical signs of infection.
  Arms: STIMULAN DEVICE USED

SUMMARY:
This is a prospective, single-center, double-blind randomized clinical trial aimed at evaluating the efficacy and safety of the extended-release antibiotic device, STIMULAN, in preventing infections in patients with open fractures. The study will enroll 40 patients from IRCSS San Raffaele's Emergency Department and Orthopedics and Traumatology Unit. Patients will be stratified into high-risk and low-risk infectious subgroups and randomized into either the intervention group receiving the antibiotic device or the control group receiving no device. The follow-up period will last for 5 days, with data collection at specified intervals. Standard laboratory tests will be utilized to monitor the patient's inflammatory response.

DETAILED DESCRIPTION:
This study is a prospective, single-center, randomized clinical trial with a double-blind design for both the patient and the evaluator. The aim is to assess the efficacy and safety of the extended-release antibiotic device STIMULAN in preventing infections in patients with open fractures.

The trial will be a randomized study that will enroll two cohorts of patients with open fractures, sourced from both the Emergency Department of IRCSS San Raffaele and the Orthopedics and Traumatology Unit. Fractures will be classified according to the Gustilo Classification. Patients requiring surgical repair of the exposed fracture will be randomized to receive either the extended-release antibiotic device or no device at all. The randomization of this study is stratified, with a 1:1 ratio, and 40 patients will be divided into two groups:

Intervention group: extended-release antibiotic device Control group: no device

Two stratification subgroups will be included:

High-risk infectious subgroup Low-risk infectious subgroup For the definition of stratification, please refer to Section 9.1, Risk Assessment Table for Stratification.

Patients will be followed for a duration of 5 days, and follow-up data will be collected at established intervals. According to recent studies, the onset of initial infections occurs between 24 and 72 hours following the episode of open fracture. Therefore, a 5-day period is deemed a reasonable time frame for constant monitoring. Standard-of-care laboratory tests such as white blood cell count, C-reactive protein, erythrocyte sedimentation rate, and procalcitonin will also be collected and analyzed to determine the patient's inflammatory response.

ELIGIBILITY:
Inclusion Criteria:

* Open fractures of any type and location
* Fractures classified as Gustilo-Anderson Type I, II, IIIa, IIIb, IIIc
* Patients requiring surgical intervention for fracture correction
* Patients with no contraindications for antibiotic treatment
* Patients providing informed consent

Exclusion Criteria:

* Patients with active infections
* Patients with a history of allergies or adverse reactions to the antibiotics used in the extended-release device
* Patients with severe renal or hepatic insufficiency
* Non-cooperative patients or those who are unable to adhere to follow-up visits or study procedures due to physical or mental limitations or severe neurological illness
* Patients who have undergone spinal surgery

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Infected Open Fracture | 5 days
  The primary outcome measure of this clinical trial is the incidence of bacterial infections following surgical intervention for open fractures in both the intervention and control arms. This will be quantified as the number of confirmed bacterial infections per total number of participants in each arm, expressed as a percentage.

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale San Raffaele, Milan, Italy